CLINICAL TRIAL: NCT01732237
Title: A Single Dose Study to Investigate the Pharmacokinetics of an Oral Microdose of JNJ-42396302, JNJ-53773187 and JNJ-42692507 in Healthy Male Subjects
Brief Title: A Study to Investigate the Pharmacokinetics of JNJ-42396302, JNJ-53773187 and JNJ-42692507 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100878; 42396302EDI1003 (Other: Janssen-Cilag International NV)
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Healthy
Keywords: Healthy; JNJ-42396302; JNJ-42692507; JNJ-53773187; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- JNJ-42396302 (Experimental): Patients will receive JNJ-42396302 100 micrograms as a single oral dose after an overnight fast of at least 10 hours.
  Interventions: Drug: JNJ-42396302
- JNJ-42692507 (Experimental): Patients will receive JNJ-42692507 100 micrograms as a single oral dose after an overnight fast of at least 10 hours.
  Interventions: Drug: JNJ-42692507
- JNJ-53773187 (Experimental): Patients will receive JNJ-53773187 100 micrograms as a single oral dose after an overnight fast of at least 10 hours.
  Interventions: Drug: JNJ-53773187

INTERVENTIONS:
Drug: JNJ-42396302 — A single dose of JNJ-42396302 100 micrograms (1 mL) will be administered orally with 240-mL non-carbonated water.
  Arms: JNJ-42396302
Drug: JNJ-42692507 — A single dose of JNJ-42692507 100 micrograms (1 mL) will be administered orally with 240-mL non-carbonated water.
  Arms: JNJ-42692507
Drug: JNJ-53773187 — A single dose of JNJ-53773187 100 micrograms (1 mL) will be administered orally with 240-mL non-carbonated water.
  Arms: JNJ-53773187

SUMMARY:
The purpose of the study is to investigate the pharmacokinetics (what the body does to the medication) of JNJ-42396302, JNJ-53773187 and JNJ-42692507 after administration of a single oral dose of 100 micrograms under fasted conditions in healthy male participants.

DETAILED DESCRIPTION:
This is a phase I, open-label (all people know the identity of the intervention) and parallel-group (each group of patients will be treated at the same time), randomized (the study medication is assigned by chance) study in healthy male participants, to investigate the pharmacokinetics of a single oral dose of 100 micrograms of JNJ-42396302, JNJ-53773187 or JNJ-42692507. The study consists of 3 phases, ie, screening phase (21 days prior to first dose of study medication), a treatment phase, and a follow up phase. In the treatment phase, participants will be divided into 3 treatment groups with 6 participants each, to receive a single dose of 100 micrograms of JNJ-42396302, JNJ-53773187 or JNJ-42692507 following an overnight fast of at least 10 hours. Safety evaluations for adverse events, clinical laboratory tests, physical examination, vital signs and electrocardiogram will be monitored throughout the study. The total duration of the study will be approximately 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant should be healthy male on the basis of physical examination, medical history, vital signs, electrocardiogram, the results of blood biochemistry and hematology tests and a urinalysis
* Participant must have a Body Mass Index of 18.5 to 30.0 kg/m2
* Have a blood pressure between 90 and 140 mm Hg systolic, inclusive, and no higher than 90 mm Hg diastolic
* Agrees to protocol-defined use of effective contraception

Exclusion Criteria:

* A positive human immunodeficiency virus-type 1 or type 2 test and Hepatitis A, B or C infection at screening or admission
* Participant with abnormal physical, vital or laboratory values
* Currently active cardiovascular, bronchospastic respiratory disease, dyspnea, diabetes mellitus, movement disorder and infectious disease

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma analyte concentration (Cmax) of JNJ-42396302 | 10, 20, 30, and 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, and 72 hours
Area under the plasma concentration time curve for JNJ-42396302 | 10, 20, 30, and 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, and 72 hours
Actual sampling time to reach the maximum plasma analyte concentration (tmax) of JNJ-42396302 | 10, 20, 30, and 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, and 72 hours
Apparent terminal elimination half-life of JNJ-42396302 | 10, 20, 30, and 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, and 72 hours
Maximum observed plasma analyte concentration (Cmax) of JNJ-53773187 | 10, 20, 30, and 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, and 72 hours
Area under the plasma concentration time curve for JNJ-53773187 | 10, 20, 30, and 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, and 72 hours
Actual sampling time to reach the maximum plasma analyte concentration (tmax) of JNJ-53773187 | 10, 20, 30, and 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, and 72 hours
Apparent terminal elimination half-life of JNJ-53773187 | 10, 20, 30, and 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, and 72 hours
Maximum observed plasma analyte concentration (Cmax) of JNJ-42692507 | 10, 20, 30, and 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, and 72 hours
Area under the plasma concentration time curve for JNJ-42692507 | 10, 20, 30, and 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, and 72 hours
Actual sampling time to reach the maximum plasma analyte concentration (tmax) of JNJ-42692507 | 10, 20, 30, and 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, and 72 hours
Apparent terminal elimination half-life of JNJ-42692507 | 10, 20, 30, and 45 minutes; 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, and 72 hours

SECONDARY OUTCOMES:
Number of patients with adverse events | within 7 days after the last dose of the study medication

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV